CLINICAL TRIAL: NCT00322153
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Memantine in Patients With Moderate-to-Severe Dementia of the Alzheimer's Type
Brief Title: A Study of the Safety and Efficacy of Memantine in Moderate to Severe Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Stephen M Graham, PhD, Senior Director, Clinical Development, Neurology, Forest Research Institute, a subsidiary of Forest Laboratories, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEM-MD-50
Record Dates: First submitted 2006-05-03; First posted 2006-05-05 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-08

CONDITIONS: Dementia of the Alzheimer's Type
Keywords: memantine; Alzheimer's disease; moderate to severe Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Oral administration, once daily.
  Interventions: Drug: Placebo
- Memantine ER (Active Comparator): 28mg, once daily. Oral administration for 24 weeks.
  Interventions: Drug: memantine ER

INTERVENTIONS:
Drug: memantine ER — 28mg(7mg capsules) once daily and oral administration for 24 weeks.
  Other Names: Namenda XR
  Arms: Memantine ER
Drug: Placebo — Matching placebo oral administration once daily.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, and efficacy of memantine compared to placebo in outpatients diagnosed with moderate-to-severe dementia of the Alzheimer's type on a concurrent acetylcholinesterase inhibitor (AChEI).

DETAILED DESCRIPTION:
Memantine is a therapeutic agent that represents a unique class of Alzheimer's disease (AD) treatment options. A once daily (QD) dosing regimen in an AD population would simplify administration for the caregiver. The purpose of this study is to evaluate the safety and efficacy of modified release memantine taken once daily in outpatients with moderate-to-severe AD on a concurrent AChEI.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients aged >/= 50 years
* Diagnostic evidence of probable Alzheimer's disease consistent with criteria from the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) and the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)
* Confirmatory magnetic resonance imaging (MRI) or computed tomographic (CT) scan within the prior 12 months.
* Mini-Mental State Examination (MMSE) scores >/= 3 and </= 14 at Screening (Visit 1) and Baseline (Visit 2)
* Ongoing daily acetylcholinesterase inhibitor (AChEI) therapy at a stable dose for at least 3 months prior to Screening (Visit 1). It is preferred that patients continue to receive the same AChEI therapy for the duration of the study.

Exclusion Criteria:

* Patients with a modified Hachinski Ischemia Score greater than 4 at Screening.
* Patients who have taken memantine within one month of Screening (Visit 1)
* Patients who have a known hypersensitivity to memantine, neramexane, rimantadine, or amantadine.
* Patients whose AChEI therapy is likely to be interrupted or discontinued during the course of the study.
* Patients who are receiving therapy with more than one AChEI.
* Patients with computed tomography (CT) or magnetic resonance imaging (MRI) evidence of hydrocephalus, stroke, a space-occupying lesion, cerebral infection, or any clinically significant central nervous system disease other than Alzheimer's disease.
* Patients with a DSM-IV Axis I disorder other than Alzheimer's disease, including amnestic disorders, schizophrenia or schizoaffective disorder, bipolar disorder, current major depressive episode, psychosis, panic, or post-traumatic stress disorder.
* Patients who, in the clinician's judgement, are likely to be placed in a nursing home within the next 6 months.
* Patients who had evidence of other neurological disorders that included, but were not limited to, stroke, Parkinson's disease, seizure disorder, or head injury with loss of consciousness within the prior 5 years
* Patients who had dementia that was complicated by other organic disease
* Patients who had dementia complicated by the presence of predominant delusions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2005-06; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Graham, PhD, Study Director — Forest Laboratories
Locations (83):
- United States (38):
  - Forest Investigative Site 010, Phoenix, Arizona
  - Forest Investigative Site 062, Costa Mesa, California
  - Forest Investigative Site 050, Fresno, California
  - Forest Investigative Site 024, San Francisco, California
  - Forest Investigative Site 071, Santa Ana, California
  - Forest Investigative Site 002, Denver, Colorado
  - Forest Investigative Site 021, Boca Raton, Florida
  - Forest Investigative Site 052, Boynton Beach, Florida
  - Forest Investigative Site 070, Delray Beach, Florida
  - Forest Investigative Site 065, Fort Myers, Florida
  - Forest Investigative Site 043, Hallandale, Florida
  - Forest Investigative Site 044, Hallandale, Florida
  - Forest Investigative Site 001, Miami, Florida
  - Forest Investigative Site 034, North Miami, Florida
  - Forest Investigative Site 068, Orlando, Florida
  - Forest Investigative Site 038, Palm Beach Gardens, Florida
  - Forest Investigative Site 008, St. Petersburg, Florida
  - Forest Investigative Site 028, Tampa, Florida
  - Forest Investigative Site 009, Snellville, Georgia
  - Forest Investigative Site 069, Joliet, Illinois
  - Forest Investigative Site 045, Kalamazoo, Michigan
  - Forest Investigative Site 014, Saint Loius, Missouri
  - Forest Investigative Site 064, Long Branch, New Jersey
  - Forest Investigative Site 011, Morristown, New Jersey
  - Forest Investigative Site 003, New Brunswick, New Jersey
  - Forest Investigative Site 048, Albany, New York
  - Forest Investigative Site 006, Buffalo, New York
  - Forest Investigative Site 004, White Plains, New York
  - Forest Investigative Site 027, Centerville, Ohio
  - Forest Investigative Site 012, Toledo, Ohio
  - Forest Investigative Site 020, Portland, Oregon
  - Forest Investigative Site 032, Greensburg, Pennsylvania
  - Forest Investigative Site 018, Jenkintown, Pennsylvania
  - Forest Investigative Site 067, East Providence, Rhode Island
  - Forest Investigative Site 041, Austin, Texas
  - Forest Investigative Site 017, San Antonio, Texas
  - Forest Investigative Site 013, Richmond, Virginia
  - Forest Investigative Site 026, Tacoma, Washington
- Argentina (23):
  - Forest Investigative Site 103, Banfield, Buenos Aires
  - Forest Investigative Site 102, Buenos Aires, Buenos Aires
  - Forest Investigative Site 118, Buenos Aires, Buenos Aires
  - Forest Investigative Site 109, Buenos Aires, Buenos Aires
  - Forest Investigative Site 104, Buenos Aires, Buenos Aires
  - Forest Investigative Site 108, Buenos Aires, Buenos Aires
  - Forest Investigative Site 114, Buenos Aires, Buenos Aires
  - Forest Investigative Site 106, Buenos Aires, Buenos Aires
  - Forest Investigative Site 119, Buenos Aires, Buenos Aires
  - Forest Investigative Site 122, Buenos Aires, Buenos Aires
  - Forest Investigative Site 107, Buenos Aires, Buenos Aires
  - Forest Investigative Site 111, Buenos Aires, Buenos Aires
  - Forest Investigative Site 121, Buenos Aires, Buenos Aires
  - Forest Investigative Site 115, Buenos Aires, Buenos Aires
  - Forest Investigative Site 116, Buenos Aires, Buenos Aires
  - Forest Investigative Site 105, La Plata, Buenos Aires
  - Forest Investigative Site 123, Lanús, Buenos Aires
  - Forest Investigative Site 112, Córdoba, Córdoba Province
  - Forest Investigative Site 124, Córdoba, Córdoba Province
  - Forest Investigative Site 110, Mendoza, Mendoza Province
  - Forest Investigative Site 125, Mendoza, Mendoza Province
  - Forest Investigative Site 113, Rosario, Santa Fe Province
  - Forest Investigative Site 120, Santa Fe, Santa Fe Province
- Chile (11):
  - Forest Investigative Site 302, Antofagasta, Antofagasta
  - Forest Investigative Site 308, Coquimbo, Elqui
  - Forest Investigative Site 301, Las Condes, Santiago Metropolitan
  - Forest Investigative Site 309, Las Condes, Santiago Metropolitan
  - Forest Investigative Site 303, Providencia, Santiago Metropolitan
  - Forest Investigative Site 310, Providencia, Santiago Metropolitan
  - Forest Investigative Site 313, Recoleta, Santiago Metropolitan
  - Forest Investigative Site 305, San Ramón, Santiago Metropolitan
  - Forest Investigative Site 304, Santiago, Santiago Metropolitan
  - Forest Investigative Site 312, Santiago, Santiago Metropolitan
  - Forest Investigative Site 306, Valdivia, Valdivia
- Mexico (11):
  - Forest Investigative Site 206, Aguascalientes, Aguascalientes
  - Forest Investigative Site 212, Saltillo, Coahuila
  - Forest Investigative Site 202, Mexico City, Federal District
  - Forest Investigative Site 207, Mexico City, Federal District
  - Forest Investigative Site 211, León, Guanajuato
  - Forest Investigative Site 205, Guadalajara, Jalisco
  - Forest Investigative Site 203, Zapopan, Jalisco
  - Forest Investigative Site 208, Monterrey, Nuevo León
  - Forest Investigative Site 204, Monterrey, Nuevo León
  - Forest Investigative Site 210, San Luis Potosí City, San Luis Potosí
  - Forest Investigative Site 213, Culiacán, Sinaloa

REFERENCES:
- [Derived] Grossberg GT, Alva G, Hendrix S, Ellison N, Kane MC, Edwards J. Memantine ER Maintains Patient Response in Moderate to Severe Alzheimer's Disease: Post Hoc Analyses From a Randomized, Controlled, Clinical Trial of Patients Treated With Cholinesterase Inhibitors. Alzheimer Dis Assoc Disord. 2018 Jul-Sep;32(3):173-178. doi: 10.1097/WAD.0000000000000261. PMID 29771687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from May 20, 2005 to April 18th, 2007 at 83 study centers in four countries (23 in Argentina, 11 in Chile, 11 in Mexico, and 38 in the US)
Pre-assignment Details: Study consisted of 1-2 weeks single-blind placebo treatment followed by 24 weeks double-blind treatment. At the end of single-blind placebo treatment, patients meeting entry criteria were randomized (1:1) to 1 of 2 double-blind treatment groups receiving memantine or placebo.
Groups:
- Placebo: Matching placebo oral administration once daily for 24 weeks.
- Memantine ER: 28mg once daily oral administration for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Memantine ER
Started | 335 (Randomized to placebo) | 342 (Randomized to Memantine ER)
SAFETY POPULATION | 335 (Safety population defined as all patients who took at least one dose of double-blind study drug.) | 341 (Safety population: one patient was randomized but did not receive double-blind study drug.)
Completed | 272 | 273
Not Completed | 63 | 69
Not completed — Adverse Event | 21 | 34
Not completed — Protocol Violation | 6 | 14
Not completed — Withdrawal by Subject | 18 | 10
Not completed — Lack of Efficacy | 8 | 3
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawn for other reasons | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Memantine ER | Total
Number analyzed (Participants) | 335 | 341 | 676
Age, Customized [Number; unit: participants]
  <= 64 years | 26 | 34 | 60
  65-74 years | 79 | 85 | 164
  75-84 years | 179 | 176 | 355
  >= 85 years | 51 | 46 | 97
Age Continuous [Mean (Standard Deviation); unit: years] | 76.8 (7.76) | 76.2 (8.35) | 76.5 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243 | 244 | 487
  Male | 92 | 97 | 189
Region of Enrollment [Number; unit: participants]
  United States | 85 | 93 | 178
  Argentina | 158 | 153 | 311
  Chile | 44 | 46 | 90
  Mexico | 48 | 49 | 97

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Severe Impairment Battery (SIB) at Week 24 (LOCF)
Description: The SIB was developed for the evaluation of cognitive function in patients with more advanced dementia, and evaluates the areas of memory, language, praxis, orientation, and attention. The SIB test items consist of simple, one-step commands presented with gestural cues that are repeated if necessary. The test contains 51 items, and the range of possible scores is 0 to 100 (with 0 being the worst result). The SIB has been shown to be a valid and reliable instrument sensitive to longitudinal change.
Time Frame: Baseline to week 24
Population: Primary efficacy analysis was based on the Intent-to-Treat (ITT) Population. The ITT Population was consisted of all patients in the Safety Population who completed at least one post-Baseline efficacy assessment in SIB or CIBIC-Plus. The last-observation-carried-forward approach was used to impute missing post-Baseline values.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Memantine ER
Number analyzed (Participants) | 327 | 332
Units on a scale | -0.4 (0.65) | 2.2 (0.65)
Statistical Analysis 1: Comparison: Placebo vs Memantine ER; The co-primary efficacy parameter was change from Baseline to Week 24 in SIB total score. Missing SIB total scores at Week 24 were imputed using the last-observation-carried-forward (LOCF) approach; Test type: Superiority or Other; p = 0.001, ANCOVA; Least-squares mean (-0.4 in placebo and 2.2 in memantine ER) are controlled for center and adjusted for SIB baseline value; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [1.0 to 4.2]

2. Primary Outcome: Clinician's Interview-Based Impression of Change With Caregiver Input (CIBIC-plus) at Week 24 (LOCF)
Description: The CIBIC-Plus is a measure of an overall clinical effect and is based on a comprehensive evaluation at Baseline and later visits of four domains: general (overall clinical status), functional (including activities of daily living), cognitive, and behavioral. A skilled clinician interviews the patient, and includes information supplied by a knowledgeable caregiver. The CIBIC-Plus is a rating of the patient's global status relative to Baseline, ranging from a score of 1, indicating "marked improvement" to a score of 4, indicating "no change" to a score of 7, indicating "marked worsening."
Time Frame: Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Memantine ER
Number analyzed (Participants) | 328 | 333
Units on a scale | 4.1 (0.07) | 3.8 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Memantine ER; The co-primary efficacy parameter was CIBIC-Plus total score at week 24. Missing CIBIC-Plus total scores at Week 24 were imputed using the last-observation-carried-forward (LOCF) approach; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline in the 19-Item Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL19) Scale at Week 24 (LOCF)
Description: The ADCS-ADL19 modified inventory consists of 19 items used to measure the functional capabilities of patients with moderate to severe dementia. Each activity-of-daily-living (ADL) item comprises a series of hierarchical subquestions ranging from the highest level of independent performance to complete loss of ability to perform the ADL Inventory. The inventory is performed by interviewing a person in close contact with the patient and covers the most usual and consistent performance of the patient over the preceding 4 weeks. Response range is 0 (total disability) to 54 (total independence).
Time Frame: Baseline to week 24
Population: The secondary efficacy analysis was based on the ITT Population. The last-observation-carried-forward approach was used to impute missing post-Baseline values.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Memantine ER
Number analyzed (Participants) | 328 | 331
Units on a scale | -1.7 (0.44) | -1.0 (0.44)
Statistical Analysis 1: Comparison: Placebo vs Memantine ER; The secondary efficacy parameter was change from Baseline at Week 24 in the total score of the 19-Item Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (ADCS-ADL19). Missing scores at week 24 were imputed using the last-observation-carried-forward (LOCF) approach; Test type: Superiority or Other; p = 0.177, ANCOVA; Least-squares mean (-1.7 in placebo and -1.0 in memantine ER) are controlled for center and adjusted for ADCS-ADL19 baseline value; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.3 to 1.8]

ADVERSE EVENTS:
Time Frame: Occurring on or after the date of the first dose of double-blind study medication and within 30 days of the date of last dose of double-blind study medication.
Arm/Group | Placebo | Memantine ER
Serious Adverse Events (participants affected / at risk) | 21/335 | 28/341
Other Adverse Events (participants affected / at risk) | 70/335 | 67/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=335) | Memantine ER (N=341)
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 3 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Rectal Prolapse (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 2
Lobar Pneumonia (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Myoclonus (Nervous system disorders) | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Excessive skin (Skin and subcutaneous tissue disorders) | 0 | 1
Proctocolectomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=335) | Memantine ER (N=341)
Fall (Injury, poisoning and procedural complications) | 26 | 19 — Treatment emergent adverse event
Urinary tract infection (Infections and infestations) | 24 | 19 — Treatment emergent adverse event
Headache (Nervous system disorders) | 17 | 19 — Treatment emergent adverse event
Diarrhoea (Gastrointestinal disorders) | 13 | 17 — Treatment emergent adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 90 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential info. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in pub. On sponsor's request, PI shall delay submission for any pub while sponsor files patent apps. If trial is multi-center, PI agrees that first publication shall be a multi-center pub.